CLINICAL TRIAL: NCT01695317
Title: Effect of Acetyl-L-carnitine in Migraine - a Randomized, Double-blind Placebo Controlled Study
Brief Title: Effect of Acetyl-L-carnitine in Migraine
Acronym: ALCAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-001624-36
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-02

CONDITIONS: Migraine
Keywords: Migraine; Preventive medication
MeSH Terms: conditions — Migraine Disorders | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetyl-L-carnitine (Active Comparator): Acetyl-L-carnitine tablets
  Interventions: Drug: Acetyl-L-carnitine
- Sugar pills (Placebo Comparator): Glucose with lemon acid
  Interventions: Drug: Acetyl-L-carnitine

INTERVENTIONS:
Drug: Acetyl-L-carnitine — Week 1: 500 mg x 3, Week 2-12: 500 mg x 6
  Other Names: ALCAR

SUMMARY:
Traditionally, beta blockers have been used for migraine prophylaxis, but in later years also antiepileptic drugs. Contraindications and side effects have to some degree limited their use, and new prophylactics that can be used by most migraine sufferers and with little side effects are in demand. One product that may seem to fulfill these requirements is Acetyl-L-carnitine, which is a dietary supplement and naturally occurs in plants and animals. L-carnitine is necessary for fatty-acid metabolism and energy production.

To our knowledge, no placebo-controlled studies have previously evaluated the efficacy of Acetyl-L-carnitine in adults with migraine.

The aims of the present study is to evaluate the efficacy of Acetyl-L-carnitine as a prophylaxis in migraine patients

DETAILED DESCRIPTION:
The study will be a single-centre double-blinded, randomized, placebo controlled crossover study with Acetyl-L-carnitine or placebo. We plan to include 72 patients. The follow up duration will be 36 weeks. The study will be performed according to Good Clinical Practice, and relying partly on the International Headache Society Guidelines for controlled trials of drugs in migraine from 2012 and partly on the guidelines divulged by the International Headache Society task force on trial guidelines for chronic migraine.

After a screening visit including a neurological consultation, eligible patients will sign an informed consent declaration before they enter a 4 week run-in (baseline) period when they keep a headache diary. After 4 weeks they return for the second visit. If they have had 2 or more migraine attacks they are allowed to proceed in the study. If they have less than 2 migraine attacks (required for proceeding in the study), they are allowed to extend the baseline period another 4 weeks. Those who then during the whole 8 week period have on average 2 or more migraine attacks per month are also allowed to proceed. Otherwise they are excluded from the study.

Details of the treatment period The duration of each of the two treatment periods is 12 weeks. During each period there will be one telephone contact at the start of each treatment period to remind patients to start with medicines, and one after 2 weeks to check compliance and side effects. In the second last week of every treatment period there will be a doctor and nurse visit with drug accounting and dispensing of new medicines for the next period. At this visit one will ensure that the patient has just enough medicines left to finish the period before the wash-out. As recommended in crossover studies, the participants enter a washout period of 4 weeks between the two treatment periods, to reduce the risk of carryover effect.

Randomization Randomization will be generated using a computerized procedure. A randomization list containing 72 patient numbers is made before the start of the study, and the patient number is then indicated on a package with medicines for that patient. The study has a crossover design, and the two different treatment periods (active or placebo) can arise to two different treatment sequences (AP or PA). Patients are therefore randomized in blocks of 4 where one of these two treatment sequences is assigned to each patient in random order. With 72 patients to be included, this means that 18 patients are randomized in each block. In each block, 50% patients have the treatment sequence AP, and 50% PA in a random order.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Signed informed consent
* Migraine with or without aura according to International Classification of Headache Disorders, second version (ICHD-2) criteria
* chronic migraine according to the ICHD-2 criteria (revision 1)
* Retrospectively have 2 or more migraine attacks per month during the last 3 month
* During the baseline period have 2 or more migraine attacks
* Debut of migraine at least one year prior to inclusion
* Start of migraine before age 50 years
* Body mass index (BMI )between 18-35 kg/m2
* No medication overuse during the last 3 months defined as headache >14 days/month combined with overuse simple analgesics >14 days/month or triptans or combined medications ≥ 10 days/month.

Exclusion Criteria:

* Interval headache not distinguishable from migraine
* Chronic tension-type headache or other headache than migraine occurring on ≥ 15 days/month with or without medication overuse
* Pregnancy, nursing or inability to use contraceptives
* Hypersensitivity to active substance
* History of angioneurotic edema, diabetes mellitus, significant psychiatric illness and/or Hospital anxiety and Depression Scale( HADS) anxiety score ≥ 11 or HADS depression score ≥ 11, and/or use of selective serotonin reuptake inhibitors (SSRI), antipsychotic medication, or antidepressant medication during the last 3 months
* Use of daily migraine prophylactics less than 3 months prior to start of study
* Previous use of Acetyl-L-carnitine
* BMI <18 kg/m2 or BMI > 35 kg/m2
* Having tried ≥ 3 prophylactic drugs against migraine during the last 5 years
* Subjects requiring detoxification from acute medication
* Patients who consistently fail to respond to any acute migraine medication
* Patients with alcohol or illicit drug dependence; 13) Subjects with renal disease or decreased renal function
* Previous or present history of asthma or vascular disease, arterial claudication included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Knut Hagen, MD, PhD, Principal Investigator — Norwegian National Headache Centre
Locations (1):
- Norwegian National Headache Centre, Trondheim, Norway

REFERENCES:
- [Result] Hagen K, Brenner E, Linde M, Gravdahl GB, Tronvik EA, Engstrom M, Sonnewald U, Helde G, Stovner LJ, Sand T. Acetyl-l-carnitine versus placebo for migraine prophylaxis: A randomized, triple-blind, crossover study. Cephalalgia. 2015 Oct;35(11):987-95. doi: 10.1177/0333102414566817. Epub 2015 Jan 19. PMID 25601916

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetyl-L-carnitine First, Then Sugar Pills: Period 1: Acetyl-L-carnitine tablets Week 1: 500 mg x 3 (1.5 g), Week 2-12: 500 mg x 6 (3.0 g) Period 2: Sugar tablets (500 mg dextrose and citric acid): Week 1: 1 tablet x 3 (1,5 g), week 2-12: 6 tablets (3.0 g)
- Sugar Pills First, Then Acetyl-L-carnitine: Period 1:
  Sugar tablets (500 mg dextrose and citric acid): Week 1: 1 tablet x 3 (1,5 g), week 2-12: 6 tablets (3.0 g) Period 2: Acetyl-L-carnitine: Week 1: 500 mg x 3 (1.5 g), Week 2-12: 500 mg x 6 (3.0 g)
Period: Period 1 in the Cross-over Design
Arm/Group | Acetyl-L-carnitine First, Then Sugar Pills | Sugar Pills First, Then Acetyl-L-carnitine
Started | 36 | 36
Completed | 34 | 35
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: Cross-over to Period 2
Arm/Group | Acetyl-L-carnitine First, Then Sugar Pills | Sugar Pills First, Then Acetyl-L-carnitine
Started | 34 | 35
Completed | 30 | 1
Not Completed | 4 | 34
Not completed — Withdrawal by Subject | 4 | 34

BASELINE CHARACTERISTICS:
Groups:
- Acetyl-L-carnitine First, Then Sugar Pills: Period 1: Acetyl-L-carnitine tablets Acetyl-L-carnitine: Week 1: 500 mg x 3, Week 2-12: 500 mg x 6
  Period 2: Glucose with lemon acid Sugar pills Week 1: 500 mg x 3, Week 2-12: 500 mg x 6
- Sugar Pills First, Then Acetyl-L-carnitine: Period 1: Glucose with lemon acid Sugar pills Week 1: 500 mg x 3, Week 2-12: 500 mg x 6
  Period 2: Acetyl-L-carnitine tablets Acetyl-L-carnitine: Week 1: 500 mg x 3, Week 2-12: 500 mg x 6
- Total: Total of all reporting groups
Arm/Group | Acetyl-L-carnitine First, Then Sugar Pills | Sugar Pills First, Then Acetyl-L-carnitine | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (14) | 39 (14) | 39 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  Norway | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Headache Days
Description: The number of days per 4 weeks with moderate or severe headache lasting ≥ 4 hours or if treated with the patient's usual headache medication (usually a triptan) as the primary endpoint.
Time Frame: last 4 weeks
Population: Headache days per four week
Measure: Mean (Standard Deviation); unit: Headache days per 4 weeks
Arm/Group | Acetyl-L-carnitine | Sugar Pills
Number analyzed (Participants) | 72 | 72
Headache days per 4 weeks | 5.1 (2.8) | 5.2 (3.3)

2. Secondary Outcome: Days With Migraine and Side Effects
Description: Secondary measures will be: Days with migraine; days with headache; hours with headache; headache intensity (0-3 scale) on days with headache; doses of analgesics; doses of triptans; days with sick leave; number of responders (≥ 50% decrease in migraine days compared with baseline); incidence of side effects recorded openly.
Time Frame: Last 4 weeks
Population: Headache hours per 4 weeks
Measure: Mean (Standard Deviation); unit: Headache hours per 4 weeks
Arm/Group | Acetyl-L-carnitine | Sugar Pills
Number analyzed (Participants) | 72 | 72
Headache hours per 4 weeks | 36.4 (30.2) | 37.0 (38.9)

ADVERSE EVENTS:
Groups:
- Sugar Pills: Glucose with lemon acid
  Sugar tablets (500 mg dextrose and citric acid): Week 1: 1 tablet x 3 (1,5 g), week 2-12: 6 tablets (3.0 g):
Arm/Group | Acetyl-L-carnitine | Sugar Pills
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 25/72 | 24/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetyl-L-carnitine (N=72) | Sugar Pills (N=72)
advedrse events (Gastrointestinal disorders) | 12 (12) | 19 (19) — Pain and/or flatulence
More severe headache (Nervous system disorders) | 6 (6) | 3 (3)
Bad taste (Nervous system disorders) | 7 (7) | 2 (2) — Bad taste of tablets

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes